CLINICAL TRIAL: NCT03302494
Title: WAveCrest Vs. Watchman TranssEptal LAA Closure to REduce AF-Mediated STroke 2. A Prospective, Multicenter, Randomized, Active Controlled, Clinical Trial of the Coherex WaveCrest® Left Atrial Appendage Occlusion System Compared to the Watchman® LAA Closure Device for the Reduction in Risk of Ischemic Stroke or Systemic Embolism in Subjects With Non-valvular Atrial Fibrillation That Have an Appropriate Rationale to Seek a Non-pharmacologic Alternative to Chronic Oral Anticoagulation.
Brief Title: WAveCrest Vs. Watchman TranssEptal LAA Closure to REduce AF-Mediated STroke 2
Acronym: WAVECREST2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed due to device design modification
Sponsor: Coherex Medical (Industry)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHX_IP014
Record Dates: First submitted 2017-09-29; First posted 2017-10-05 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Non-valvular Atrial Fibrillation; Left Atrial Appendage
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: If the subject is suspected of having a stroke since their most recent follow-up, a Neurologist blinded to subject's randomization and implanted device must evaluate the subject or otherwise provide rationale for why an in-person neurology visit and exam are unnecessary. Neurology or blinded trial personnel should also administer mRS & NIHSS if there is suspicion of stroke A Clinical Events Committee, also blinded to subject's randomization, will adjudicate primary safety and effectiveness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- WaveCrest (Experimental): WaveCrest left atrial appendage occluder
  Interventions: Device: Coherex WaveCrest® Left Atrial Appendage Occlusion System
- Watchman (control) (Active Comparator): Watchman left atrial appendage closure device
  Interventions: Device: Watchman® LAA Closure Device

INTERVENTIONS:
Device: Coherex WaveCrest® Left Atrial Appendage Occlusion System — Percutaneous left atrial appendage closure
  Arms: WaveCrest
Device: Watchman® LAA Closure Device — Percutaeous left atrial appendage closure
  Arms: Watchman (control)

SUMMARY:
The WAVECREST 2 trial is a prospective, multicenter, randomized, active controlled, clinical trial to evaluate the safety and effectiveness of the Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System.

DETAILED DESCRIPTION:
The WAVECREST 2 trial is a prospective, multicenter, randomized, active controlled, clinical trial to evaluate the safety and effectiveness of the Coherex WaveCrest Left Atrial Appendage (LAA) Occlusion System. Subjects will be randomized in a 1:1 ratio to the Treatment Arm (Coherex WaveCrest LAA occlusion system) or the Control Arm (Boston Scientific's Watchman LAA occlusion system). The trial is designed to demonstrate that safety and effectiveness of the WaveCrest device are non-inferior to the Watchman device.

ELIGIBILITY:
Inclusion Criteria:

1. Documented evidence of paroxysmal, persistent, or permanent non-valvular atrial fibrillation
2. At least 18 years of age
3. Calculated CHADS2 score ≥ 2 or CHA2DS2-VASc score ≥ 3
4. Indication for warfarin therapy with an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulation
5. Willing and able to comply with post-implant anticoagulation and antiplatelet regimen
6. Willing to participate in the required follow-up visits and tests
7. Subject has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the IRB/EC at the site

Exclusion Criteria:

1. Atrial fibrillation (AF) due to a reversible cause (e.g. thyrotoxicosis or postoperative)
2. Known contraindication and/or allergy to warfarin, nickel, aspirin, intravenous contrast or P2Y12 inhibitors (clopidogrel, ticagrelor, and prasugrel), which cannot be adequately pre-medicated or desensitized
3. Conditions other than AF requiring long-term anticoagulation therapy
4. Contraindications for percutaneous catheterization procedures
5. Prior surgical LAA occlusion/exclusion or implanted with LAA occlusion device, or any prior attempt of such procedures
6. Prior percutaneous or surgical closure of a patent foramen ovale or atrial septal defect
7. Inability or unwillingness to take oral anticoagulation for 45 days post-procedure
8. New York Heart Association (NYHA) Class IV heart failure
9. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant
10. History of symptomatic carotid, intervertebral, or intracranial artery occlusion or stenosis without revascularization with the exception of known occlusion without symptoms > 6 months
11. Modified Rankin Scale (mRS) score ≥ 4
12. Chronic resting heart rate ≥ 110 bpm
13. Congenital cardiac anomalies requiring cardiac surgery or interventional repair
14. Stroke or transient ischemic attack (confirmed by Neurologist) within 60 days prior to enrollment
15. Myocardial infarction within 60 days prior to enrollment
16. Sepsis or any infection requiring oral antibiotic therapy within 14 days or intravenous antibiotic therapy within 30 days prior to enrollment
17. Surgical or interventional cardiovascular and non-cardiovascular procedure including cardioversion within 30 days prior to enrollment or AF ablation within 60 days prior to enrollment or any planned general surgery or interventional procedure within 90 days after enrollment or any planned cardiac surgery.
18. On renal replacement therapy, serum creatinine > 3.0 mg/dl (265 μmol/L) or calculated creatinine clearance < 25 ml/minute
19. Thrombocytopenia (<60,000 platelets/mm3), leucopenia (white blood cell count < 3,000 cells/mm³), or anemia (hemoglobin concentration < 10 grams/deciliter) based on blood work done within 30 days prior to enrollment
20. Any medical disorder or psychiatric illness that would interfere with successful completion of the trial
21. Currently participating in an investigational drug trial or another device trial that has not completed the primary endpoint (trials requiring extended follow-up for products that are commercially available are not considered investigational trials). Concurrent enrollment in the ACC LAAO Registry is permitted.
22. Subject belongs to a vulnerable population (see definition in Appendix I: Acronyms and Definitions)
23. Any condition that would reduce life expectancy to less than 2 years
24. Women of childbearing potential who are, or plan to become pregnant during the time of the trial (method of assessment per physician discretion)

Echocardiographic Exclusion Criteria

1. Left ventricular ejection fraction < 30%
2. Mitral valve stenosis defined as valve area < 1.5cm2, mean gradient > 6mmHg, or any valve deformity consistent with rheumatic valvular disease
3. Aortic valve stenosis defined as valve area ≤1.0cm2 or mean gradient >30mmHg
4. Circumferential pericardial effusion > 10mm or symptomatic pericardial effusion
5. Evidence of intracardiac thrombus
6. Cardiac tumor or myxoma
7. Atrial septal defect that warrants closure
8. Complex atheroma in the ascending aorta or aortic arch as evidenced by mobile plaque
9. Left Atrial Appendage size and shape are unsuitable for closure with a WaveCrest or Watchman device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Study Chair — MOUNT SINAI HOSPITAL; Gregg Stone, MD, Study Chair — MOUNT SINAI HOSPITAL
Locations (25):
- United States (23):
  - Grandview Medical Center, Birmingham, Alabama
  - Dignity Health Mercy Gilbert Medical Center, Chandler, Arizona
  - Pacific Heart Institute / St. John's Health Center, Los Angeles, California
  - Medstar Heart and Vascular Institute - Washington Hospital Center, Washington D.C., District of Columbia
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Wellstar Kennestone, Marietta, Georgia
  - Baptist Health Lexington, Lexington, Kentucky
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Marquette General Hospital, Marquette, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Northwell Health, Bay Shore, New York
  - New York University- NYU Langone Cardiac, New York, New York
  - New York University, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University, Columbus, Ohio
  - UPMC Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Heart Hospital Baylor Plano (Baylor Research Institute), Plano, Texas
  - Christus Trinity Clinic Research, Tyler, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Monash Health, Melbourne
  - St. Vincent's Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analysis population included participants greater than or equal to (>=) 18 years old diagnosed with non-valvular atrial fibrillation and a CHADS2 score >= 2 or a CHA2DS2-VASc score >= 3 who had an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulation.
Pre-assignment Details: As pre-specified in the protocol, participants who signed the informed consent form (ICF) were considered enrolled in the study. Out of the 248 enrolled participants (who signed the ICF), 183 were randomized to respective treatment arms, 26 were screen failures and 39 discontinued due to study hold during the screening period. Hence, data for 183 randomized participants is reported below.
Groups:
- Group 1 (WaveCrest Roll-In): Roll in participants who were enrolled prior to a site's randomization phase and who had vascular access attempted, underwent Coherex WaveCrest left atrial appendage (LAA) occlusion system (WaveCrest device) implant procedure. Coherex Wave Crest LAA occlusion system delivery sheath was used to deliver the implant percutaneously via the femoral vein through a transseptal puncture into the LAA.
- Group 2 (WaveCrest Randomized): Randomized participants underwent Coherex WaveCrest LAA occlusion system (WaveCrest device) implant procedure. Coherex Wave Crest LAA occlusion system delivery sheath was used to deliver the implant percutaneously via the femoral vein through a trans septal puncture into the LAA.
- Group 3 (Watchman Randomized): Randomized participants underwent Watchman left atrial appendage closure (LAAC) System (Watchman Device) implant procedure. Watchman device was intended for percutaneous, transcatheter closure of the left atrial appendage and consisted of the watchman access system (access sheath and dilator) and watchman delivery system (delivery catheter and watchman device). The access sheath and delivery catheter permitted device placement in the LAA via femoral venous access and inter-atrial septum crossing into the left atrium.
Period: Overall Study
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
Started | 71 | 54 | 58
Treated | 71 | 52 | 56
Completed | 6 | 1 | 3
Not Completed | 65 | 53 | 55
Not completed — Other | 7 | 4 | 6
Not completed — Withdrawal by Subject | 10 | 2 | 9
Not completed — Study Terminated by Sponsor | 32 | 29 | 30
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 3
Not completed — Death | 13 | 11 | 4
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Randomized but not treated and discontinued during study hold | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (mITT) analysis set consisted of all randomized participants who had vascular access attempted for the implant procedure of the intended left atrial appendage (LAA) occlusion device.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized) | Total
Number analyzed (Participants) | 71 | 52 | 56 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (9.64) | 75.9 (6.43) | 76.0 (5.69) | 74.4 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 21 | 20 | 73
  Male | 39 | 31 | 36 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 69 | 51 | 53 | 173
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of All Cause Death, Procedure or Device Related Complications Requiring Percutaneous or Surgical Intervention or Major Bleeding
Description: The primary safety outcome was the composite of death from any cause (all-cause mortality), procedure or device related complications requiring percutaneous or surgical intervention through 45 days post procedure or major bleeding throughout the duration of the trial. The analysis was based on sponsor assessment of adverse events data. Baseline was defined as 90 day prior to treatment or 90 days prior to randomization; baseline assessments could occur on the day of implant.
Time Frame: All death, procedure- or device-related complications requiring percutaneous or surgical intervention: From baseline up to 45 days; major bleeding: From baseline up to 5 years 11 months
Population: The intention-to-treat (ITT) analysis set consisted of all randomized participants regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
Number analyzed (Participants) | 71 | 52 | 56
Percentage of participants | 47.89 [35.9 to 60.1] | 32.69 [20.3 to 47.1] | 17.86 [8.9 to 30.4]

2. Primary Outcome: Percentage of Participants With Composite of Ischemic Stroke or Systemic Embolism at 24 Months
Description: Percentage of participants with composite of ischemic stroke or systemic embolism at 24 months was reported.
Time Frame: At 24 months
Population: The ITT analysis set consisted of all randomized participants regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
Number analyzed (Participants) | 71 | 52 | 56
Percentage of participants | 4.23 [0.9 to 11.9] | 3.85 [0.5 to 13.2] | 5.36 [1.1 to 14.9]

3. Secondary Outcome: Percentage of Participants With Ischemic Stroke or Systemic Embolism With the WAVECREST Device in Comparison to the CHADS2 and CHA2DS2-VASc Imputed Risk of Ischemic Stroke or Systemic Embolism in the Absence of Anticoagulant Therapy
Description: CHADS2 (congestive heart failure, hypertension, age >=75 years (yrs), prior Stroke/transient ischemic attack (TIA)/Thromboembolism) and CHA2DS2-VASc scores (Vascular disease, Age 65- 74 yrs, female Sex) were developed to identify non-valvular atrial fibrillation (AF) participants at an elevated risk for ischemic stroke. CHADS2 score assign 1 point: congestive heart failure, hypertension, age >= 75 yrs, diabetes mellitus; 2 points: prior stroke/TIA/thromboembolism. CHADS2 score ranges from 0 to 6. Higher scores indicated higher risk for ischemic strokes. CHA2DS2-VASc Score assign 1 point for each following risk factors: congestive heart failure, hypertension (blood pressure consistently above 140/90), diabetes mellitus, vascular disease, age 65 to74 yrs, female and assigned 2 points for age >=75 yrs and prior stroke or TIA or thromboembolism each. Overall score ranged from 0 to a 9, with lower scores indicated lower risk and higher scores indicated higher risk for ischemic strokes.
Time Frame: At 45 days
Population: The ITT analysis set consisted of all randomized participants regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
Number analyzed (Participants) | 71 | 52 | 56
Percentage of participants
  ischemic strokes | 4.23 | 3.85 | 5.36
  systemic embolisms | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Left Atrial Appendage (LAA) Closure
Description: Percentage of participants with LAA closure, defined as a gap of <= 5 millimetre (mm) at the 45-day visit as assessed by transesophageal echocardiogram (TEE) was reported.
Time Frame: At 45 days
Population: Analysis population included all roll-in and randomized and treated participants. Here 'N' (number of participants analysed) signifies number of participants who were evaluable for this outcome measures.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1 (WaveCrest Roll-In) | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
Number analyzed (Participants) | 67 | 50 | 51
Percentage of participants | 100.0 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Baseline up to 5 years 11 months
Description: ITT analysis set consisted of all randomized participants regardless of treatment received.
Groups:
- Group 1 (WaveCrest Roll-In):: Roll in participants who were enrolled prior to a site's randomization phase and who had vascular access attempted, underwent Coherex WaveCrest left atrial appendage (LAA) occlusion system (WaveCrest device) implant procedure. Coherex Wave Crest LAA occlusion system delivery sheath was used to deliver the implant percutaneously via the femoral vein through a transseptal puncture into the LAA.
Arm/Group | Group 1 (WaveCrest Roll-In): | Group 2 (WaveCrest Randomized) | Group 3 (Watchman Randomized)
All-Cause Mortality (participants affected / at risk) | 15/71 | 13/52 | 4/56
Serious Adverse Events (participants affected / at risk) | 50/71 | 42/52 | 39/56
Other Adverse Events (participants affected / at risk) | 63/71 | 51/52 | 48/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (WaveCrest Roll-In): (N=71) | Group 2 (WaveCrest Randomized) (N=52) | Group 3 (Watchman Randomized) (N=56)
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 3
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 11 | 7 | 5
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 4 | 2 | 4
Cardiac failure congestive (Cardiac disorders) | 6 | 6 | 6
Cardiac tamponade (Cardiac disorders) | 2 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 2 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 4 | 0 | 0
Pericardial effusion (Cardiac disorders) | 9 | 2 | 1
Pericarditis (Cardiac disorders) | 2 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 4 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
leus (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Asthenia (General disorders) | 2 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 5 | 2 | 2
Death (General disorders) | 1 | 1 | 1
Device embolisation (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 1
Medical device site thrombosis (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 3
Corona virus infection (Infections and infestations) | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 2 | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 1
Influenza (Infections and infestations) | 0 | 2 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 6 | 6
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 5 | 2 | 3
Septic shock (Infections and infestations) | 2 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 3
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection fraction abnormal (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Paracentesis (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 2
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 1
Dementia (Nervous system disorders) | 0 | 2 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 3 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Mixed dementia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 2
Visual field defect (Nervous system disorders) | 1 | 0 | 0
Wernicke's encephalopathy (Nervous system disorders) | 1 | 0 | 0
Device defective (Product Issues) | 1 | 0 | 0
Device leakage (Product Issues) | 1 | 0 | 0
Device loosening (Product Issues) | 0 | 0 | 1
Device malfunction (Product Issues) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 3 | 2 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 2
Haematoma (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (WaveCrest Roll-In): (N=71) | Group 2 (WaveCrest Randomized) (N=52) | Group 3 (Watchman Randomized) (N=56)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 6
Atrial fibrillation (Cardiac disorders) | 13 | 8 | 4
Pericardial effusion (Cardiac disorders) | 11 | 12 | 12
Eye disorders (Eye disorders) | 8 | 1 | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 15 | 10 | 13
Chest pain (General disorders) | 8 | 5 | 7
Fatigue (General disorders) | 2 | 3 | 4
Oedema peripheral (General disorders) | 6 | 3 | 6
Cellulitis (Infections and infestations) | 4 | 4 | 3
Corona virus infection (Infections and infestations) | 9 | 9 | 5
Urinary tract infection (Infections and infestations) | 10 | 5 | 9
Contusion (Injury, poisoning and procedural complications) | 7 | 2 | 4
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 4
Laceration (Injury, poisoning and procedural complications) | 8 | 5 | 5
Investigations (Investigations) | 8 | 4 | 6
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 14 | 13 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 6
Dizziness (Nervous system disorders) | 4 | 4 | 4
Syncope (Nervous system disorders) | 3 | 3 | 3
Psychiatric disorders (Nervous system disorders) | 5 | 1 | 4
Acute kidney injury (Renal and urinary disorders) | 9 | 2 | 6
Haematuria (Renal and urinary disorders) | 3 | 4 | 7
Reproductive system and breast disorders (Reproductive system and breast disorders) | 4 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 11 | 4 | 5
Hypertension (Vascular disorders) | 1 | 6 | 3
Hypotension (Vascular disorders) | 7 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this clinical study may be submitted for publication without regard for whether the trial results are positive or negative. Sponsor will be responsible for oversight of the publication process and will have oversight of publications of results of the trial, the Physician Advisory Committee may advise.

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03302494/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT03302494/SAP_001.pdf